CLINICAL TRIAL: NCT02497066
Title: Randomized, Controlled, Double-blind, Efficacy Study Comparing Compounded Topical Pain Creams vs. Placebo for Treating Pain Symptoms
Brief Title: Efficacy Study Comparing Compounded Topical Pain Creams vs. Placebo for Treating Pain Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #412770-2
Record Dates: First submitted 2015-06-30; First posted 2015-07-14 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2018-10

CONDITIONS: Pain
Keywords: topical; compound; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neuropathic Pain (Placebo Comparator): Subjects with neuropathic pain will receive a neuropathic pain cream combined of Ketamine 10%/Gabapentin 6%/Clonidine 0.2% and Lidocaine 2% or placebo. They will be told to use the pain cream 3 times per day. Each will receive cream in identical dispensers. Cream is dispensed by rotating the base of the device and each rotation also produces a clicking sound. The number of clicks will be standardized so that all doctors utilize the same prescription depending on the size of the patient's pain location.
  Interventions: Other: Neuropathic pain cream
- Nociceptive pain (Placebo Comparator): Subjects with nociceptive pain will receive a nociceptive pain cream combined of Ketoprofen 10%/Baclofen 2%/Cyclobenzaprine 2% and Lidocaine 2% or placebo. They will be told to use the pain cream 3 times per day. Each will receive cream in identical dispensers. Cream is dispensed by rotating the base of the device and each rotation also produces a clicking sound. The number of clicks will be standardized so that all doctors utilize the same prescription depending on the size of the patient's pain location.
  Interventions: Other: Nociceptive pain cream
- Mixed pain (Placebo Comparator): Subjects who have a mixed (nociceptive and neuropathic) pain conditions will receive a mixed pain cream combined of Ketamine 10%/Gabapentin 6%/Diclofenac 3%/baclofen 2%/Cyclobenzaprine 2% and Lidocaine 2% or placebo. They will be told to use the pain cream 3 times per day. Each will receive cream in identical dispensers. Cream is dispensed by rotating the base of the device and each rotation also produces a clicking sound. The number of clicks will be standardized so that all doctors utilize the same prescription depending on the size of the patient's pain location.
  Interventions: Other: Mixed pain cream

INTERVENTIONS:
Other: Neuropathic pain cream — Subjects will apply the cream to the painful area.
  Arms: Neuropathic Pain
Other: Nociceptive pain cream — Subjects will apply the cream to the painful area.
  Arms: Nociceptive pain
Other: Mixed pain cream — Subjects will apply the cream to the painful area.
  Arms: Mixed pain

SUMMARY:
The main objective of this protocol is to determine the effectiveness of using compounded topical pain creams for treating neuropathic, nociceptive, or mixed-pain syndromes. Since these compounded pain creams may be associated with burning or irritation at the application site, and possible systemic effects may present, the secondary objective is to determine the relative satisfaction with the creams. The investigators hypothesis is that the active pain creams may provide significant benefit compared to placebo cream.

3.1 Specific Aims

1. Specific Aim 1 will determine pain relief following treatment with the appropriate (based on specified pain) compounded topical pain cream or a placebo cream. The investigators hypothesis is that the compounded topical pain creams will provide greater pain relief than placebo creams.
2. Specific Aim 2 will measure the patient satisfaction with the cream (compound or placebo). The investigators hypothesis is that the compounded topical pain creams will improve patient satisfaction, while the placebo cream will not result in a change in patient satisfaction with their pain treatment.

DETAILED DESCRIPTION:
In this study, the investigators are attempting to determine whether compounded topical pain creams are more effective than placebo; as well as measuring the subjects' satisfaction with the compounded pain creams. Three different compounded pain creams (specific to the type of pain being treated) will be used to examine effectiveness and satisfaction in treating neuropathic, nociceptive, or mixed pain syndromes. Up to 399 subjects will be randomized to receive a compounded pain cream or placebo. The type of pain cream to be used will be based on the subjects' pain diagnosis. Pain relief will be measured by a 0-10 Numeric Rating Scale and satisfaction by a 1-5 Likert Satisfaction Scale. The outcome measures will include a 'positive outcome' defined as a two point or greater reduction in average pain (as measured by a NRS) and a score of greater than 3 (on a 1-5 Likert scale measuring satisfaction) at 1-month. The investigators will use the Rand Corporation SF-36 to measure changes in health status during enrollment. Subjects who obtain benefit at 1-month will be followed at 3-months, while those who fail to obtain benefit (i.e., ≥ 2 point reduction in NRS with a greater than 3 Likert satisfaction score) will exit the study to receive alternative care. Patients will be given a pain diary so that their NRS can be calculated at follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18;-90
2. A localized pain complaint to include: the back, neck, face, groin, buttocks, abdomen, chest, or up to two extremities
3. Average pain score ≥ 4/10 over the past week;
4. Pain duration > 6 weeks
5. DEERS eligibility.

Exclusion Criteria:

1. Previous prescription for a compounded pain cream.
2. Cannot read or understand English.
3. Allergic reaction to Ketamine, Gabapentin, Diclofenac, Baclofen, Cyclobenzaprine, Ketoprofen, Clonidine or lidocaine.
4. Pregnancy. Ruling out pregnancy will be done in accordance with our standard procedures, which is to obtain a urine HCG in any female of child-bearing age who may be pregnant prior to starting any new medications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) 0-10 | 1 month
  The Numerical Pain Rating Scale is a unidimensional measure of pain intensity. It is an 11 point numerical scale (with 0 meaning no pain; and 10 meaning the worst possible pain imaginable) used to assess pain intensity for persons able to self-report.

SECONDARY OUTCOMES:
Change in Health Status via Rand Corporation SF-36 | 1 month
  The SF-36 is a 36 item Short Form Health Survey that is used to measure changes in health status. It is a set of generic, coherent, and easily administered quality-of-life measures. It is a validated measure of 8 domains including emotional health and physical function, with lower scores translating to greater disability.
5-point Likert Satisfaction Scale (1-5) | 1 month
  The 5-point Likert Satisfaction Scale is a 5 point scale that is used to measure the subjects opinion/perception of their satisfaction with the compounded product. The scale ranges from 1-5; with 1 denoting "very unsatisfied" and 5 signifying "very satisfied."
Composite outcome determined by combining the subjects average change in pain score measured by the Numerical Pain Rating Scale and their score on the 5-point Likert Satisfaction Scale. | 1 month
  A positive composite outcome was defined as a decrease in average pain of 2 points or greater and a satisfaction score greater than 3.
Numerical Pain Rating Scale (NPRS) 0-10 | 3 months
  The Numerical Pain Rating Scale is a unidimensional measure of pain intensity. It is an 11 point numerical scale (with 0 meaning no pain; and 10 meaning the worst possible pain imaginable) used to assess pain intensity for persons able to self-report.
Change in Health Status via Rand Corporation SF-36 | 3 Months
  The SF-36 is a 36 item Short Form Health Survey that is used to measure changes in health status. It is a set of generic, coherent, and easily administered quality-of-life measures. It is a validated measure of 8 domains including emotional health and physical function, with lower scores translating to greater disability.
5-point Likert Satisfaction Scale (1-5) | 3 months
  The 5-point Likert Satisfaction Scale is a 5 point scale that is used to measure the subjects opinion/perception of their satisfaction with the compounded product. The scale ranges from 1-5; with 1 denoting "very unsatisfied" and 5 signifying "very satisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Brutcher, PharmD,Ph.D., Principal Investigator — WRNMMC

REFERENCES:
- [Derived] Brutcher RE, Kurihara C, Bicket MC, Moussavian-Yousefi P, Reece DE, Solomon LM, Griffith SR, Jamison DE, Cohen SP. Compounded Topical Pain Creams to Treat Localized Chronic Pain: A Randomized Controlled Trial. Ann Intern Med. 2019 Mar 5;170(5):309-318. doi: 10.7326/M18-2736. Epub 2019 Feb 5. PMID 30716769